CLINICAL TRIAL: NCT02295176
Title: Metabolic and Cardiovascular Effects of a Proprietary Nutraceutical Containing Berberine, Policosanols and Red Yeast in Subjects With Metabolic Syndrome
Brief Title: Metabolic and Cardiovascular Effects of Armolipid Plus in Subjects With Metabolic Syndrome
Acronym: ARMP-11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rottapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARMP-11
Record Dates: First submitted 2014-11-05; First posted 2014-11-20 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Metabolic Syndrome; Insulin-resistance; Left Ventricular Hypertrophy
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Hypertrophy, Left Ventricular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armolipid Plus (Experimental): Armolipid Plus: 1 tablet daily in the evening after dinner for 24 weeks.
  Interventions: Dietary Supplement: Armolipid Plus
- Placebo (Placebo Comparator): 1 tablet matching Armolipid Plus daily in the evening after dinner for 24 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Armolipid Plus
  Arms: Armolipid Plus
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Aim of the study is to evaluate the effects of Armolipid Plus on insulin sensitivity in patients with MetS and increased LV mass.

168 patients will be enrolled in this randomized, double-blind, parallel-group, placebo-controlled trial and treated for 24 weeks.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a highly prevalent condition characterized by visceral obesity, abnormalities of glucidic and lipid metabolism, and increased risk for cardiovascular events. Such findings appear to be associated with a decrease in insulin sensitivity. Management of metabolic syndrome is currently aimed at treating individual components of the disease without addressing this underlying pathophysiologic mechanism; this translates into multidrug regimens, high costs and patient compliance issues.

A complication of hypertension is hypertrophy of the left ventricle (LV), which is closely related to the incidence of cardiovascular events whose regression results in a proportional reduction of the risk. But also other factors contribute as sex, age, race, genetics, diet and insulin resistance.

MetS is closely related to hypertrophy of the LV. Therefore it is possible that the treatment of MetS may be an effective strategy for the prevention of organ damage.

Armolipid Plus (an association of berberine 500mg, red yeast rice titled in 3 mg monacolin K,- policosanol 10 mg, coenzyme Q10 2mg,astaxanthin 0,5mg, folic acid 0,2mg) has been found to be effective at reducing blood cholesterol and triglycerides, and at improving endothelial function; subgroup analyses also suggested a benefit on glucose metabolism, myocardial mass and improved diastolic function in subjects with MetS and early organ damage.

Aim of the study is to evaluate the effects of Armolipid Plus on insulin sensitivity in patients with MetS and increased LV mass.

168 patients will be enrolled in this randomized, double-blind, parallel-group, placebo-controlled trial; active treatment will consist of Armolipid Plus (1 tbl qd).

Primary end point will be the reduction of the insulin resistance in patients with metabolic syndrome and increased LV mass.

ELIGIBILITY:
Inclusion Criteria:

* male and Female 18-70 aged, with diagnosis of metabolic syndrome, defined by the presence of waist circumference >102 cm (♂) or >88 cm(♀), and two or more of these criteria:

  * fasting blood glucose >100 mg
  * systolic blood pressure >135 or diastolic blood pressure >85 mmHg or patients in treatment with antihypertensive drugs
  * triglyceridemia >150 mg/dl
  * HDL cholesterolemia < 40 mg/dl(M), < 50 mg/dl(F).
* left ventricular hypertrophy: left ventricular mass indexed to height >44 g/m2,7(♀)or >48 g/m2(♂).
* antihypertensive and lipid-lowering therapy (if applicaple) stable for at least three months.
* ability to understand and sign an informed consent form.

Exclusion Criteria:

* pregnancy or lactation period
* diabetes mellitus or pharmacological treatment for this condition
* hepatic failure
* creatininemia >2mg/dl
* triglyceridemia >500mg/dl
* severe obesity (BMI >35)
* chronic renal failure with glomerular filtration rate <30ml/min
* triglycerides >500mg/dl
* left ventricular systolic dysfunction (LVEF <40%)
* hypertrophic cardiomyopathy
* valvular stenosis
* previous myocardial infarction with acinesie
* intermediate or severe cardiac valve disorders
* intolerance to any components of Armolipid Plus
* pacemaker generated arrhythmia
* Inadequately controlled high blood pressure during therapy optimization (SBP >140mmHg or DBP >90mmHg)
* patients with comorbidities are allowed (e.g. ischemic heart disease, dysthyroidism) but they have got to be in stable therapy for at least 3 months and they did not have major clinical events in the last three months;
* heart failure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure will be the reduction of the insulin/glucose ratio, both after overnight fast (HOMA index) | 6 months

SECONDARY OUTCOMES:
cardiac remodeling assessed by echocardiogram, lipid profile, subtypes of LDL, blood pressure, and high-sensitivity C-reactive protein. | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Domenico Bonaduce, Naples, Naples
  - Ferruccio Galletti, Naples
  - Giuseppe Schillaci, Terni

REFERENCES:
- [Derived] Mercurio V, Pucci G, Bosso G, Fazio V, Battista F, Iannuzzi A, Brambilla N, Vitalini C, D'Amato M, Giacovelli G, Vaudo G, Schillaci G, Galletti F, Bonaduce D. A nutraceutical combination reduces left ventricular mass in subjects with metabolic syndrome and left ventricular hypertrophy: A multicenter, randomized, double-blind, placebo-controlled trial. Clin Nutr. 2020 May;39(5):1379-1384. doi: 10.1016/j.clnu.2019.06.026. Epub 2019 Jul 19. PMID 31371114